CLINICAL TRIAL: NCT05464888
Title: Animal Assisted Therapy's Effects on Young Dental Patients
Brief Title: Animal Assisted Therapy in Pediatric Dentistry
Acronym: AAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1454
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- +Short AAT (Experimental): Children aged 4-8 y.o. willing to receive an oral exam, a toothbrush cleaning, simulated radiographs and be a study participant - 75 experimental patients who will be interacting with the dog prior to their oral exam.
  Interventions: Behavioral: +Short AAT
- +Long AAT (Experimental): Children aged 4-8 y.o. willing to receive an oral exam, a toothbrush cleaning, simulated radiographs and be a study participant - 75 experimental patients who will be interacting with the dog throughout their entire visit.
  Interventions: Behavioral: +Long AAT
- Active control; NO dog (Active Comparator): Children aged 4-8 y.o. willing to receive an oral exam, a toothbrush cleaning, simulated radiographs and be a study participant - 75 control patients who will not be interacting with the dog during their visit and will color a dog picture for 3 minutes instead.
  Interventions: Behavioral: Active control; NO dog

INTERVENTIONS:
Behavioral: +Short AAT — Interaction with therapy dog prior to dental exam, cleaning, and simulated radiographs.
  Arms: +Short AAT
Behavioral: +Long AAT — Interaction with therapy dog throughout dental exam, cleaning, and simulated radiographs.
  Arms: +Long AAT
Behavioral: Active control; NO dog — Color dog picture for 3 minutes prior to dental exam, cleaning, and simulated radiographs.
  Arms: Active control; NO dog

SUMMARY:
A prospective randomized trial measuring physiologic biometrics and perceptions of stress during a pediatric dental exam, cleaning, and simulated radiographs with or without a therapy dog present.

DETAILED DESCRIPTION:
Patients will be consented, enrolled, and randomly assigned to a control group (no dog) or to an experimental group with dog present only before their dental visit for 3 minutes (+ Short AAT) or to an experimental group with dog present throughout their entire visit (+ Long AAT). Control (no dog) patients will have an active control where they color for 3 minutes before their dental exam, cleaning, and simulated radiographs, without a dog present. Biometric data will be collected with a small wireless wrist device (Shimmer 3) which measures heart rate and sweat response (skin galvanic response). Salivary samples will be taken before and after the dental visit to measure salivary cortisol and amylase, as a metric of physiological stress. Finally, a video feed of body movements during the dental visit will be collected for observational coding. Pre-visit and post-visit surveys will be given to all the patients on their experiences regarding pain, anxiety, and perceptions of the dental experience.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

* 4-8 years of age
* English speaking
* Qualifies for a dental exam and prophylaxis (cleaning) by having not received a dental prophylaxis or oral exam in the past 3 months
* Stable physical health, decided at the discretion of the study coordinator and PI
* Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based on research site personnel's assessment
* Evidence of a personally signed and dated informed assent form from the child and legal guardian's consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial and all of their questions have been answered

Exclusion Criteria: Subjects presenting with any of the following will not be included in the study:

* Patients <4yo and >8yo
* Non-English speakers
* Patients unwilling to assent/participate or parental/guardian consent was not given
* Self-report or parental report of patient suffering current dental pain
* Known allergies or significant adverse reactions following exposure to dogs or the use of oral hygiene products (toothpastes, mouth rinses), and all ingredients in prophy paste
* Children who are afraid of dogs or had a prior negative experience with dogs as reported by the parent or child
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this trial
* Developmental/cognitive disability such that patient cannot self-assent, comprehend and follow the requirements of the study based on research site personnel's assessment

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean Heart Rate during Dental Exam | During dental exam, approximately 2- 5 minutes.
  Beats per minute during dental exam. Heart rate measured using wrist-worn Shimmer heart rate tracking device.
Mean Heart Rate during Dental Cleaning | During dental cleaning, approximately 2- 5 minutes.
  Beats per minute during dental cleaning. Heart rate measured using wrist-worn Shimmer heart rate tracking device.
Mean Heart Rate during Dental Radiograph Simulation | During dental radiograph simulation, approximately 2- 5 minutes.
  Beats per minute during dental radiograph simulation. Heart rate measured using wrist-worn Shimmer heart rate tracking device.
Salivary Cortisol during Dental Exam | During dental exam, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.
Salivary Cortisol during Dental Cleaning | During dental cleaning, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.
Salivary Cortisol during Dental Radiograph Simulation | During dental radiograph simulation, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.
Salivary Amylase during Dental Exam | During dental exam, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.
Salivary Amylase during Dental Cleaning | During dental cleaning, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.
Salivary Amylase during Dental Radiograph Simulation | During dental radiograph simulation, approximately 1-2 minutes.
  To measure stress levels salivette swab will be placed in child's cheek to absorb saliva. Swabs are spun down for extraction and saliva sample will undergo ELISA assay to measure cortisol level.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Jacox, DMD, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- General & Oral Health Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 to 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Kapov G, Linton K, Gatewood C, Liu C, Strauman T, Hodges E, Graves C, Sawicki C, Wu D, Divaris K, Jacox LA. Effects of animal-assisted therapy on dental anxiety, behavior, and perceptions in young pediatric patients: a blinded randomized controlled trial. Trials. 2025 Aug 7;26(1):279. doi: 10.1186/s13063-025-08970-z. PMID 40775655